CLINICAL TRIAL: NCT05762666
Title: Pain Monitoring in Intensive Care: How the Use of Nociception Level Index Affects Treatment and Prognosis?
Brief Title: Nociception Level Index as Monitorization of Pain at the Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 212-2022
Record Dates: First submitted 2023-01-11; First posted 2023-03-09 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Intensive Care, Surgical; Anesthesia, General
Keywords: nociception level index; Postoperative pain; behavioral pain scores; pain monitoring; delirium; postoperative cognitive dysfunction
MeSH Terms: conditions — Pain, Postoperative; Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Intervention Model Description: Group A will be followed with standard monitorization only along with pain scales and receive rescue analgesia according to them. However, Group B will acquire NOL monitorization throughout the ICU stay and have the same rescue analgesia under NOL guidance with concurrent pain scales.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Data obtained at the clinical follow-up will be gathered by care provider nurses at the ICU who are blind to the study protocol. All evaluations at the surgical wards especially for delirium and cognitive dysfunction will be evaluated by the same independent anesthetist who is blind to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Standart of care (No Intervention): Patients will be followed with standard monitorization only along with pain scales and receive rescue analgesia according to them
- Group Nociception level index monitor (Experimental): Patients will acquire NOL monitorization throughout the ICU stay and have the same rescue analgesia under NOL guidance with concurrent pain scales
  Interventions: Device: nociception level index monitor

INTERVENTIONS:
Device: nociception level index monitor — The nociception level index (NOL) is one of the new electrophysiological devices to asses pain-related nociception and differs with its multi-parameter evaluation. It is generated from five different parameters (heart rate, heart rate variability, skin conductance level, photo-plethysmography waveform amplitude, number of skin conductance fluctuations, and their time derivatives)
  Arms: Group Nociception level index monitor

SUMMARY:
The aim of our study is to evaluate the effectiveness of a nociception monitor in providing adequate postoperative analgesia for patients needing critical care after surgery. Besides, the study searches to determine the difference between the amount of analgesic medication used when guided by nociception or standard pain management protocols. It is also aimed to reveal the incidence of delirium when pain management is managed under the nociception level index (NOL) guidance.

60 postoperative patients admitted to the postanesthesia care unit (PACU) after general anesthesia for surgery for more than 2 hours will be included and allocated into 2 groups(n=30): the control group (Group A) and the study group (Group B). Group Standard of care will be followed with standard monitorization only along with pain scales and receive rescue analgesia according to them. However, Group NOL will acquire NOL monitorization throughout the ICU stay and have the same rescue analgesia under NOL guidance with concurrent pain scales. Data to be recorded are total postoperative analgesic consumption, NOL values along with CPOT scores, and delirium.

DETAILED DESCRIPTION:
the investigators designed a prospective study after approval of our Institutional ethics committee (dossier no:212-2022) and planned to allocate 60 patients (2 groups; 1:1 allocation; n=30). This study is designed under the Declaration of Helsinki and written informed consent will be obtained before surgery. Patients within the study should have general anesthesia for surgery for more than 2 hours and also planned for follow-up at the postanesthesia care unit (PACU). Among these, an investigator selects patients aged over 18 and having American society of anesthesiology (ASA) scores I-III. Exclusion criteria are refusal to participate in the study; patients with additional organ failure especially lung failure (Pao2/fio2 value below 200); history of allergies to drugs used in the study protocol; patients receiving deep anesthesia with sedation infusion RASS -2 (unable to be awakened by uncooperative audible stimulus); patients with head trauma expected to have a low postoperative Glasgow coma score (GCS); the presence of surgical complication, arrhythmia, and sepsis during the hospital stay.

Randomization is designed with concealed opaque envelope in a 1:1 ratio into 2 groups (n= 30): the control group (Group Standard of care) and the study group (Group NOL). When the inclusion/exclusion criteria are met, on the day of the surgery the anesthetist in the operating room will choose one envelope to apply the designed protocol for each group. Data obtained at the clinical follow-up will be gathered by informed nurses at the ICU. All evaluations at the surgical wards especially for delirium and cognitive dysfunction will be evaluated by the same independent anesthetist who is blind to the study groups.

All patients will receive standard analgesia protocol as 1 gr paracetamol (maximum dose 4x1 and minimum dose interval as 6 hours) and rescue analgesia as 1mg/kg tramadol (maximum dose 4x1 and minimum dose interval as 6 hours). Moreover, if analgesia is not ensured 0,05 mg/kg morphine (IV) bolus doses are planned when their pain scales or NOL values are high (NRS >4; CPOT>2; NOL >25 over 1 minute). NRS and CPOT will be used as pain scales at postoperative 6th, 8th, 12th, and 24th hours for all patients. The Group Standard will be followed with standard monitorization only along with pain scales and receive rescue analgesia according to them. However, Group NOL will acquire NOL monitorization throughout the ICU stay and have the same rescue analgesia under NOL guidance with concurrent pain scales. The total amount of analgesics used during the ICU stay will be noted. Delirium and cognitive dysfunction will be evaluated at the 24th hour before discharge by CAM-ICU score and by 4AT at the surgical ward on the postoperative 3rd day before hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status classification I to III
* Patients who have been admitted to the postoperative intensive care unit
* Patients necessitating general anesthesia for surgery of more than 2 hours
* Patients who need mechanical ventilation for a while in intensive care follow-up

Exclusion Criteria:

* Patients with additional organ failure
* Disease that may make it difficult to wean from the ventilator when lung functions are evaluated (Pao2/fio2 value below 200)
* History of allergies to drugs used in the study protocol
* Patients receiving deep anesthesia with sedation infusion RASS -2 (unable to be awakened by uncooperative audible stimulus)
* Patients with head trauma expected to have a low postoperative Glasgow coma score
* Presence of arrhythmia
* Presence of sepsis during the hospital stay
* Patients who stay more than 48 hours at the postoperative intensive care unit
* Presence of surgical complication
* Known hepatic insufficiency or decreased function
* Known renal insufficiency or decreased function

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
critical care observation pain tool | postoperative 24 hour
  critical care observation pain tool (CPOT) behavioral pain assessment score over 2 is accepted as pain to apply analgesia
number rating scale(NRS) | postoperative 24 hour
  number rating scale(NRS) value over 4 is accepted as pain to apply analgesia

SECONDARY OUTCOMES:
The total amount of analgesic drug | postoperative 24 hour
  morphine and tramadol used at postoperative follow-up
Delirium | postoperative 24th hour
  Confusion Assessment Method for the ICU (CAM-ICU) at 24th hour : outcome will be decided as positive or negative after interrogation of course of mental status, consciousness, inattention and disorganized thinking
cognitive dysfunction | postoperative 24th hour and postoperative 3th day
  Arousal, Attention, Abbreviated Mental Test (4AT) scores at 24th hour and postoperative 3th day: A score of 1-3 suggests cognitive impairment and a score of 4 or more suggests delirium

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelinas C, Shahiri T S, Richard-Lalonde M, Laporta D, Morin JF, Boitor M, Ferland CE, Bourgault P, Richebe P. Exploration of a Multi-Parameter Technology for Pain Assessment in Postoperative Patients After Cardiac Surgery in the Intensive Care Unit: The Nociception Level Index (NOL)TM. J Pain Res. 2021 Dec 7;14:3723-3731. doi: 10.2147/JPR.S332845. eCollection 2021. PMID 34908872
- [Result] Chanques G, Gelinas C. Monitoring pain in the intensive care unit (ICU). Intensive Care Med. 2022 Oct;48(10):1508-1511. doi: 10.1007/s00134-022-06807-w. Epub 2022 Jul 29. No abstract available. PMID 35904563
- [Result] Kotfis K, van Diem-Zaal I, Williams Roberson S, Sietnicki M, van den Boogaard M, Shehabi Y, Ely EW. The future of intensive care: delirium should no longer be an issue. Crit Care. 2022 Jul 5;26(1):200. doi: 10.1186/s13054-022-04077-y. PMID 35790979